CLINICAL TRIAL: NCT01326169
Title: ReDIAL: A Telephone Brief Intervention for Injured Emergency Department Patients
Acronym: ReDIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Michael J. Mello, MD, MPH, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AA017895 (NIH)
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Alcohol Drinking
Keywords: Alcohol; brief intervention; injuries
MeSH Terms: conditions — Alcohol Drinking; Wounds and Injuries | interventions — Crisis Intervention; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Standard care (Active Comparator): No intervention
  Interventions: Behavioral: Standard care
- Counseling (Experimental): Telephone-delivered counseling
  Interventions: Behavioral: Brief intervention

INTERVENTIONS:
Behavioral: Brief intervention — Telephone-delivered counseling
  Arms: Counseling
Behavioral: Standard care — No intervention
  Arms: Standard care

SUMMARY:
The goal of this study is to reduce impaired driving, risky driving and alcohol-related negative consequences among injured emergency department (ED) patients through a telephone brief intervention. This study will allow researchers to test a novel method of brief intervention that has the potential to be convenient and efficient mechanism to deliver an intervention to an at-risk population. Eligible patients will be consented in the ED, will receive an assessment and then will be randomized into one of two conditions: 1) telephone brief intervention or 2) a comparison control group with a home safety educational program. The participant will also receive an appointment for an initial telephone call. Both conditions will be provided over three telephone sessions: the initial call (immediately following randomization) and two booster calls at 2 weeks and 6 weeks after randomization. Participants will provide information about their alcohol use, alcohol-related injuries, impaired driving, and other driving related negative consequences at 4, 8, and 12 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Age greater than 17 years
* ASSIST score >=11
* Injured Emergency Department patient at time of consent

Exclusion Criteria:

* Medically unable to give consent
* Not English or Spanish speaking
* Homeless
* Cannot be contacted by telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in number of patients with alcohol-related negative consequences from baseline to 4, 8, and 12 months post-randomization | Change from baseline in alcohol-related negatve consequences at 4, 8, and 12 months
  Specifically, the effect of the intervention on alcohol-related injuries and alcohol-related psychosocial consequences from baseline at 4, 8, and 12 months post-randomization.

SECONDARY OUTCOMES:
Evaluation of mechanisms of change model | 12 months post-randomization
  Determine the moderators and mediators of primary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mello, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Mello MJ, Baird J, Lee C, Strezsak V, French MT, Longabaugh R. A Randomized Controlled Trial of a Telephone Intervention for Alcohol Misuse With Injured Emergency Department Patients. Ann Emerg Med. 2016 Feb;67(2):263-75. doi: 10.1016/j.annemergmed.2015.09.021. Epub 2015 Nov 14. PMID 26585044